CLINICAL TRIAL: NCT03682887
Title: Cryoballoon Pulmonary Vein Isolation vs. Cryoballoon Pulmonary Vein Isolation With Additional Right Atrial Linear Ablation for Persistent Atrial Fibrillation: Prospective Randomized Trial (CRARAL Trial)
Brief Title: Cryoballoon Pulmonary Vein Isolation vs. Cryoballoon Pulmonary Vein Isolation With Additional Right Atrial Linear Ablation for Persistent Atrial Fibrillation (CRARAL Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0734
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Cryoballoon; Linear ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Sample Size Determination A. 276 subjects will be enrolled in this study. After enrollment, subjects will be randomized in a 1:1 fashion to Cryoballoon PV isolation group (138 subjects) or Cryoballoon PV isolation group with additional RA linear ablation group (138 subjects).
  B. The difference in the recurrence of atrial fibrillation between the two groups will be identified based on the data, with 80% statistical power and a 5% two-sided alpha error rate, to examine the 16% estimated difference between the groups, considering an about 5% dropout rate. The clinical recurrence rate of atrial fibrillation in the general control group was set at 39.3% considering the existing literature and the data of this hospital.
  C. Statistical hypothesis: There is a significant difference in the clinical recurrence and risk of complications after cryoballoon pulmonary vein isolation and additional right atrial linear ablation for persistent atrial fibrillation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon PV isolation group (Active Comparator): 1. Pulmonary vein isolation will be performed using a cryoballoon catheter.
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. A 28mm cryoballoon catheter will be used.
  4. Cryoablation will be performed for 180 secs at -30 C or below on condition that the pulmonary vein is occluded with a cryoballoon.
  5. CMAP (compound motor action potential) monitoring will be done to avoid phrenic nerve damage during the freezing of the right superior pulmonary vein.
  6. The procedure and ablation times will be evaluated.
  7. The procedure will be completed without checking any other trigger came from beyond pulmonary vein after the administration of isoproterenol
  8. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: Cryoballoon PV isolation group
- Cryoballoon PV isolation w/ RA linear ablation group (Experimental): 1. Pulmonary vein isolation will be performed using a cryoballoon catheter as the same as cryoballoon PV isolation group.
  2. Additional cavo-tricuspid isthmus ablation will be performed with a radiofrequency catheter.
  3. Additional SVC-right atrial septal linear ablation will be performed with a radiofrequency catheter.
  4. If any other trigger came from beyond pulmonary vein is detected after the administration of isoproterenol, additional local RF ablation will be followed.
  5. The procedure and ablation times will be evaluated.
  6. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: Cryoballoon PV isolation with Additional RA linear ablation group

INTERVENTIONS:
Procedure: Cryoballoon PV isolation group — 1. Prospective randomization (cryoballoon PV isolation group vs. cryoballoon PV isolation group with additional RA linear ablation group) (Using the Python program, a random number module is imported with the import random syntax, and the random number table for the two groups is created.)
  2. Target number of subjects: 278 (138 per group)
  3. Rhythm FU : ECG during every visit (1, 3, 6, and 12 months, and then every 6 months thereafter or upon the recurrence of symptoms after AFCA) and 24-h Holter monitor recording at 3 and 6 months and every 6 months thereafter.
  4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
  5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.
  Arms: Cryoballoon PV isolation group
Procedure: Cryoballoon PV isolation with Additional RA linear ablation group — 1. Prospective randomization (cryoballoon PV isolation group vs. cryoballoon PV isolation group with additional RA linear ablation group) (Using the Python program, a random number module is imported with the import random syntax, and the random number table for the two groups is created.)
  2. Target number of subjects: 278 (138 per group)
  3. Rhythm FU : ECG during every visit (1, 3, 6, and 12 months, and then every 6 months thereafter or upon the recurrence of symptoms after AFCA) and 24-h Holter monitor recording at 3 and 6 months and every 6 months thereafter.
  4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
  5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.
  Arms: Cryoballoon PV isolation w/ RA linear ablation group

SUMMARY:
Cryoballoon ablation is proven to be effective in pulmonary vein isolation in patients with paroxysmal atrial fibrillation. However, it is not certain that cryoablation is effective and safe in patients with persistent atrial fibrillation, because of higher chance of recurrence compared to paroxysmal atrial fibrillation. The aim of this study is to evaluate the efficacy and safety of cryoballoon pulmonary vein isolation vs. cryoballoon pulmonary vein isolation with additional right atrial linear ablation for paroxysmal atrial fibrillation in a prospective randomized trial

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (cryoballoon PV isolation group vs. cryoballoon PV isolation group with additional RA linear ablation group) (Using the Python program, a random number module is imported with the import random syntax, and the random number table for the two groups is created.)
2. Target number of subjects: 278 (138 per group)
3. Rhythm FU : ECG during every visit (1, 3, 6, and 12 months, and then every 6 months thereafter or upon the recurrence of symptoms after AFCA) and 24-h Holter monitor recording at 3 and 6 months and every 6 months thereafter.
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.

Cryoballoon PV isolation group

1. Pulmonary vein isolation will be performed using a cryoballoon catheter.
2. Esophageal temperature will be monitored to prevent esophageal injury.
3. A 28mm cryoballoon catheter will be used.
4. Cryoablation will be performed for 180 secs at -30ºC or below on condition that the pulmonary vein is occluded with a cryoballoon.
5. CMAP (compound motor action potential) monitoring will be done to avoid phrenic nerve damage during the freezing of the right superior pulmonary vein.
6. The procedure and ablation times will be evaluated.
7. The procedure will be completed without checking any other trigger came from beyond pulmonary vein after the administration of isoproterenol
8. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.

Cryoballoon PV isolation with Additional RA linear ablation group

1. Pulmonary vein isolation will be performed using a cryoballoon catheter as the same as cryoballoon PV isolation group.
2. Additional cavo-tricuspid isthmus ablation will be performed with a radiofrequency catheter.
3. Additional SVC-right atrial septal linear ablation will be performed with a radiofrequency catheter.
4. If any other trigger came from beyond pulmonary vein is detected after the administration of isoproterenol, additional local RF ablation will be followed.
5. The procedure and ablation times will be evaluated.
6. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Followed up for a minimum of 12 months after ablation.
3. Outpatient clinic visits regularly at 1, 3, 6, and 12 months, and then every 6 months thereafter or upon the recurrence of symptoms after AFCA Rhythm control at 2 months, and thereafter every 6-month follow-up with
4. ECG during every visit and 24-h Holter monitor recording at 3 and 6 months and every 6 months thereafter.
5. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

C. Follow-up Patients were followed up for a minimum of 12 months after ablation. All the patients will be followed-up at 1, 3, 6, and 12 months, and thereafter every 6 months. If the patient shows any symptom within the clinical study period, patient will visit the outpatient clinic. ECG will be performed at every outpatient visits, and 24-hour Holter or event recording will be performed every 6 months for 2 years, and every year after 2 years (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines). If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed in 12-lead ECG or Holter, it will be evaluated as recurrence. Recurrence within 3 months after the procedure will be classified as early recurrence, and that after 3 months will be classified as clinical recurrence.

9. Observation Items • Clinical Test Items and Observation Method A. Disease name, age, gender, weight, height, disease duration B. Evaluation of comorbid structural heart disease pattern C. Evaluation of clinically significant comorbid disease pattern D. Imaging quantitative assessment (All the examinations will be performed according to the need for treatment, regardless of the purpose of the study, and no additional imaging tests will be performed for study purposes.)

1. Echocardiography: Ejection fraction, diastolic function index, atrial size, ventricular size, atrial volume
2. 3D CT scan: Atrial size, ventricular size, atrial volume, and pericardial fat volume (This examination is indispensable for the safety of the procedure and for the use of 3D equipment in catheter ablation for atrial fibrillation in all clinical studies. The analysis of the atrial size, pericardial fat volume, etc. will be utilized for the purpose of risk assessment for recurrence-related factor detection and future recurrence risk. In other words, the purpose is to provide better treatment for patients at a higher level.) E. Hemodynamic quantitative evaluation: Measurement of atrial pressure before and after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient with persistent atrial fibrillation who is scheduled for ablation procedure
* ≥20 and ≤80 years of age
* LA size ≤ 45mm
* Patient who is indicated for anticoagulation therapy(for prevention of cerebral infarction) and antiarrhythmic drug

Exclusion Criteria:

* Patients with paroxysmal or permanent atrial fibrillation
* Atrial fibrillation associated with severe cardiac malformation or a structural heart disease that is hemodynamically affected
* Patients with severe renal impairment or CT imaging difficulty using contrast media
* Patients with a past history of radiofrequency ablation for atrial fibrillation or other cardiac surgery
* Patients with active internal bleeding
* Patients with contraindications for anticoagulation therapy (for prevention of cerebral infarction) and antiarrhythmic drugs
* Patients with valvular atrial fibrillation (mitral stenosis >grade 2, mechanical valve)
* Patients with a severe comorbid disease
* Expected survival < 1 year
* Drug addicts or alcoholics
* Patients who cannot read the consent form (illiterates, foreigners, etc.)
* Other patients who are judged by the principal or sub-investigator to be ineligible for participation in this clinical study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence of any atrial arrhythmia | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.
  Recurrence of any atrial arrhythmia (Defined as atrial fibrillation, atrial tachycardia, or atrial flutter lasting at least 30 seconds after a 3-month post-procedure blanking period

SECONDARY OUTCOMES:
Procedure time | immediate after procedure
Anti-arrhythmic drug use after a 3-month blanking period | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.
Recurrence of any atrial arrhythmia lasting at least 30 seconds occurring after a 3-month blanking period or anti-arrhythmic drug use after a 3-months blanking period | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.
Number of patients with recurrence as atrial fibrillation | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.
Number of patients with recurrence as atrial tachycardia/flutter | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.
Procedural complications | immediate after procedure
Proportion of cardioversion performed among patients with the recurrence of atrial arrhythmia. | up to 24 months with a minimum of 12 months follow up after a single ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Nam Pak, Principal Investigator — Yonsei University Health system, Severance Hospital
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No